CLINICAL TRIAL: NCT03686904
Title: Investigating the Effect of an Anti-Biofilm Solution to Reduce Bacterial Burden and Accelerate Healing in Chronic Wounds.
Brief Title: Investigation of a Novel Wound Gel to Improve Wound Healing in Chronic Wounds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Next Science TM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0218
Record Dates: First submitted 2018-08-02; First posted 2018-09-27 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2020-01

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection | interventions — Debridement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- SOC GROUP [Cohort A] (Placebo Comparator): Debridement, SOC irrigation & SOC topical gel
  Interventions: Other: standard of care topical gel; Procedure: Debridement; Other: Saline Irrigation (SOC Irrigation)
- SOC TOPICAL GEL & TORRENT X GROUP [Cohort B] (Active Comparator): Debridement, benzalkonium irrigation & SOC topical gel
  Interventions: Other: standard of care topical gel; Procedure: Debridement; Drug: benzalkonium irrigation
- BLASTX and SALINE (SOC) GROUP [Cohort C] (Active Comparator): Debridement, SOC saline irrigation & benzalkonium gel
  Interventions: Drug: Benzalkonium Gel; Procedure: Debridement; Other: Saline Irrigation (SOC Irrigation)
- BLASTX and TORRENTX GROUP [Cohort D] (Active Comparator): Debridement, benzalkonium irrigation & benzalkonium gel
  Interventions: Drug: Benzalkonium Gel; Procedure: Debridement; Drug: benzalkonium irrigation

INTERVENTIONS:
Drug: Benzalkonium Gel — antibiofilm solution (BlastX) topical wound gel
  Other Names: BlastX
  Arms: BLASTX and SALINE (SOC) GROUP [Cohort C]; BLASTX and TORRENTX GROUP [Cohort D]
Other: standard of care topical gel — standard of care topical gel (hydrocolloid topical gel)
  Other Names: Topical Antibacterial gel
  Arms: SOC GROUP [Cohort A]; SOC TOPICAL GEL & TORRENT X GROUP [Cohort B]
Procedure: Debridement — Removing dead tissue from infected wound (in clinic)
  Other Names: local debridement
Drug: benzalkonium irrigation — washing and lavaging in clinic with benzalkonium irrigation
  Other Names: TorrentX
  Arms: BLASTX and TORRENTX GROUP [Cohort D]; SOC TOPICAL GEL & TORRENT X GROUP [Cohort B]
Other: Saline Irrigation (SOC Irrigation) — Normal Saline Irrigation (SOC Irrigation)
  Other Names: SOC Irrigation
  Arms: BLASTX and SALINE (SOC) GROUP [Cohort C]; SOC GROUP [Cohort A]

SUMMARY:
This is a prospective, randomized, double-blinded, single site study examining the impact of a biofilm-based treatment of chronic wounds of the lower extremity. 200 subjects will be enrolled in this study. Benzalkonium solution wound irrigation and Benzalkonium wound gel will be compared to standard of care wound preparation and dressing (NS wound irrigation and hydrocolloid gel) following local debridement. Wounds will be assessed maximum of 12 weeks with a minimum of 4 follow up visits. Patients will be recruited from the general wound clinic population. No enticement will be offered and participation will be completely voluntary. At enrollment and at each follow up visit the wound will be assessed for size (length, width, and depth), signs of infection or irritation, qualitative and quantitative cultures will be taken before and after debridement, patients will be assessed for compliance to the treatment protocol, satisfaction with their treatment, any adverse effects of the treatment, and hospitalizations since last assessment. It is anticipated that enrollment and completion of the study will take 1 year.

DETAILED DESCRIPTION:
The role of biofilm in causing wound infections and preventing healing is unclear. Preliminary data suggests that persistent biofilm following excisional debridement may re-inoculate clean wounds leading to infection. Additionally, this data also suggests that persistent biofilm leads to chronic wound inflammation. Novel wound gels have been developed which claim to disrupt biofilm and kill biofilm producing bacteria. Patients presenting with a chronic wound will be randomized to receive treatment with a novel anti-biofilm solution BlastX™(benzalkonium gel) or standard of care. All patients presenting with a chronic wound (>4 weeks duration) will be assessed for eligibility in the study. If eligible, subjects will be randomized into Cohort A (debridement, NS irrigation, SOC topical wound treatment), Cohort B (debridement, benzalkonium irrigation, SOC topical wound treatment), Cohort C (debridement, NS irrigation, and benzalkonium topical wound treatment) of Cohort D (debridement, benzalkonium irrigation, and benzalkonium topical wound treatment). Subjects will receive this treatment until the wound is completely healed or they are exited from the study.

Infection of chronic wounds is a multifactorial process involving the interplay between host factors, the condition of the wound, and the number and virulence of bacterial species that flourish and critically colonize in the tissue. 1 It is widely recognized that the microorganisms colonizing in these wounds are biofilm producers. 2, 3, 4, 5 Biofilm is a polymeric slime layer made up of polymeric sugars, microbial and/or host DNA, microbial proteins and host molecules that encapsulate microorganisms.5 This limits the reach of the host immune system and antibacterial agents. Biofilm formation has been associated with the emergence of a diverse group of opportunistic pathogens, such as Staphylococcus aureus and Pseudomonas aeruginosa, which contribute to recurrent infections by modifying environmental parameters.4

Excisional debridement is the standard of care for chronic wound management and has shown to be effective against biofilm. However, studies have shown that biofilm formation recurs within 24hrs of debridement. Common topical wound preparations contain silver, iodine, honey, or chlorhexidine; none of which have shown efficacy against biofilm.1 Recent studies have reported that when targeting and disrupting the wound biofilm matrix, wound healing outcomes are improved and there is a significant decrease in biofilm-related infections. 3, 5 To date, there is no widely accepted topical agent which targets biofilm.

Preliminary and invitro studies have shown benzalkonium chloride to be an effective agent to disrupt biofilm and prevent recolonization. An example of a commercially available formulation of benzalkonium chloride is Benzalkonium gel wound gel and Benzalkonium solution wound irrigation. There is insufficient clinical data suggesting whether a biofilm focused approach is superior or inferior to standard of care treatment. In order to determine the clinical efficacy of a biofilm-focused approached against current stand of care treatment, this study outlines a clinical study evaluating the outcomes of patients treated with Benzalkonium gel and Benzalkonium solution compared to standard of care wound gel and irrigation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-99
2. Chronic wound requiring debridement
3. Wound located anywhere on the body
4. Able to comply with clinical trial requirements

Exclusion Criteria:

1. Patient unable or unwilling to comply with study requirements
2. Disease or treatment causing substantial immunosuppression
3. History of allergic reaction to benzalkonium
4. Transplant recipient

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Colony Forming Units Count Measure (Primary Measure) | 12 weeks
  The primary outcome is the change in CFU counts after treatment with Benzalkonium solution/Benzalkonium gel or SOC.

SECONDARY OUTCOMES:
Change in index ulcer size measured in cm squared (Secondary endpoints) | 12 weeks
  Change in index ulcer size measured in cm squared
Duration of index ulcer measured in weeks (Secondary endpoints) | 12 weeks
  Duration of index ulcer measured in weeks

OTHER OUTCOMES:
Measurement of local perfusion using specialized noninvasive imaging (Tertiary endpoints) | 12 weeks
  We will explore the association between the treatment and change in local perfusion using hyperspectral imaging.
Measurement of time to heal subjects wounds | 12 weeks
  Interaction of time with treatment and other baseline covariates will be included and tested

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Attinger, MD, Principal Investigator — MedStar Georgetown University Hospital
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Data was not collected for use in future research and will not be shared